CLINICAL TRIAL: NCT01908686
Title: Pivotal Response Treatment for Children With Autism Spectrum Disorders
Acronym: PRT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 1106008625; 2R01NS035193-18 (NIH)
Record Dates: First submitted 2013-07-22; First posted 2013-07-26 (Estimated); Last update posted 2020-08-14 (Actual); Status verified 2020-08

CONDITIONS: Autism Spectrum Disorders
Keywords: ASD
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pivotal Response Training (Active Comparator): Pivotal Response Training with children ages 4-35 years of age with an Autism Spectrum Disorder diagnosis
  Interventions: Behavioral: Pivotal Response Training
- Waitlist Control (No Intervention): Children in WL will be offered treatment following WL condition.

INTERVENTIONS:
Behavioral: Pivotal Response Training — Behavioral intervention for autism
  Other Names: Pivotal Response Treatment
  Arms: Pivotal Response Training

SUMMARY:
The purpose of this study is to evaluate the application of an evidence-based, manualized treatment for children with Autism Spectrum Disorder (ASD) (Pivotal Response Treatment, PRT) to children ages four through six years of age with ASD. Specifically, children will be randomly assigned to receive either (1) 10 hours per week of intervention services, including two hours per week of parent education, and eight hours per week of direct clinician-delivered services, or (2) a treatment as usual control. Intervention will focus on enhancing the following developmental skills: expressive and receptive language, play, and social interaction. Outcome measures will address changes in the aforementioned domains during structured observation and standardized assessment.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria:

Participants will:

1. Fit the age requirement: age 4-35
2. Have been diagnosed previously with an ASD and meet criteria for ASD when characterized by research team.
3. Be in good medical health
4. Be cooperative with testing
5. English is a language spoken in the family
6. Successfully complete an fMRI and EEG scan
7. Full-scale IQ>50

Exclusion Criteria:

* Exclusion Criteria:

Participants may not have:

1. Any metal or electromagnetic implants, including:

   1. Cardiac pacemaker
   2. Defibrillator
   3. Artificial heart valve
   4. Aneurysm clip
   5. Cochlear implants
   6. Shrapnel
   7. Neurostimulators
   8. History of metal fragments in eyes or skin
2. Significant hearing loss or other severe sensory impairment
3. A fragile health status.
4. Current use of prescription medications that may affect cognitive processes under study.
5. A history of significant head trauma or serious brain or psychiatric illness

Ages: 4 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2012-05; Primary Completion 2019-12-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Social Responsiveness Scale (SRS) Total Score | 16 weeks

SECONDARY OUTCOMES:
Clinical Global Impressions Scale (CGI-I) | 16 weeks
Autism Diagnostic Observation Schedule (ADOS) Comparison Score | 16 weeks
Aberrant Behavior Checklist (ABC) | 16 weeks
Vineland Domain Scores | 16 weeks
Change in Eye Tracking (ET) patterns | 16 weeks
Change in neural response to social stimuli using fMRI | 16 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Yale Child Study Center - Autism Program, New Haven, Connecticut, United States